CLINICAL TRIAL: NCT03997227
Title: Erector Spinae Plane (ESP) Block For Postoperative Pain Management In Lumbar Spine Surgery : A Randomized Control Trial
Brief Title: Erector Spinae Plane (ESP) Block For Postoperative Pain Management In Lumbar Spine Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Sinan ASAR, Principal Investigator, clinical research, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019/04
Record Dates: First submitted 2019-05-27; First posted 2019-06-25 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Erector Spinae Block

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Block group (Active Comparator)
  Interventions: Procedure: Erector spinae Block
- control group (No Intervention)

INTERVENTIONS:
Procedure: Erector spinae Block — After anesthesia and surgical procedures, a bilateral ESP block with ultrasound guidance will be applied from the T10 level at the middle line 3 cm lateral. Prior to the block, with povidone iodine, the T10 transverse protrusion will be determined by using linear ultrasound probe. The local anesthetic will be applied between the transverse projection and the erector spina muscle with the help of an isolated needle designed for peripheral block operations. Without local anesthesia, the location of the needle with saline will be confirmed by hydrodissection. After confirming the location of the needle, 20 ml of LA and saline mixture will be applied and the same procedure will be repeated in the control. A total of 40 ml of LA, 20 ml of bupivacaine 0.5%, 10 ml of lidocaine 2%, 10 ml of saline will be composed of saline.
  Arms: Block group

SUMMARY:
Lumbar vertebra surgery is one of the most common surgical procedures. After lumbar veretebra surgery, patients complain of excessive pain. Postoperative pain usually occurs in the early postoperative period and delays patient mobilization and thus lengthens hospital stay.

The aim of this study was to investigate the effect of this field block on postoperative pain and respiratory function in patients undergoing ESP with lomber vertebra surgery and with ultrasound guidance for postoperative analgesia.

DETAILED DESCRIPTION:
Lumbar vertebra surgery is one of the most common surgical procedures. After lumbar veretebra surgery, patients complain of excessive pain. Postoperative pain usually occurs in the early postoperative period and delays patient mobilization and thus lengthens hospital stay.

The aim of this study was to investigate the effect of this field block on postoperative pain and respiratory function in patients undergoing ESP with lomber vertebra surgery and with ultrasound guidance for postoperative analgesia.

ASA I-III, 68 patients between 18-75 years of age were planned to be included in the study. 34 participants were expected to be included in the control and implementation group.

In our study, the ESP block was planned to be applied to the patients in the block group. Peroperative analgesia plan will be applied to all patients in the same way. In this protocol, intravenous paracetamol 1 gr and tramadol 1 mg / kg were determined. Then, every eight hours, paracetamol and contromal infusion.

At the end of the operation, the patients will be determined by the Numeric Rating Scale (NRS) system at the 30th hour, 1st, 6th, 12th and 24th hours after the first hour of the operation. Tramadol PCA and paracetamol are administered every eight hours.

Age, sex, weight, body mass index, application of ESP block, time of surgery, duration of surgery, evaluation of pain in postoperative recovery room and 24-hour follow-up will be recorded when the patient is mobilized and discharged.

It is thought that the ESP block will decrease postoperative pain by providing effective pain control after surgery in patients undergoing lumbar vertebra surgery. In addition, it is thought to accelerate mobilization in the postoperative period and shorten the time of discharge.

ELIGIBILITY:
Inclusion Criteria:

* 68 patients
* ASA I-III,
* Aged 18-75 years
* underwent lumbar spine surgery under elective conditions

Exclusion Criteria:

* Presence of contraindications to LA agents used in this study
* Use of chronic opioids,
* Psychiatric disorders.
* Surgical procedures that lasted <60 minutes or> 300 minutes
* The presence of infection at the injection area.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2019-05-02 (Actual); Primary Completion 2020-05-02 (Estimated); Study Completion 2020-07-02 (Estimated)

PRIMARY OUTCOMES:
NRS(numerical rating scala) | 24 hours
  Each item is scored 0-10 ( 0=no pain, 10= pain as bad as can be) Postoperative pain intensity reported with NRS score : 30. minute, 1. hours, 6. hours, 12. hours, 24. hours
pruritus, nausea and vomiting, use of antiemetics | 24 hours
  each criterion is reported as present or absent each criterion is reported as present or absent
mobilized , discharged | 7 days
  each criterion is reported as when the patient is mobilized and when he is discharged

CONTACTS AND LOCATIONS:
Overall Officials: Sinem Sarı, Principal Investigator — Aydin Adnan Menderes University
Locations (1):
- Adnan Menderes Univesity, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Almeida CR, Oliveira AR, Cunha P. Continuous Bilateral Erector of Spine Plane Block at T8 for Extensive Lumbar Spine Fusion Surgery: Case Report. Pain Pract. 2019 Jun;19(5):536-540. doi: 10.1111/papr.12774. Epub 2019 Mar 15. PMID 30758122